CLINICAL TRIAL: NCT07110662
Title: New Therapeutic Approach to Toxic Epidermal Necrolysis (TEN) Using Anti-CD38+ Antibodies in the Active Phase of the Disease - Phase I/II Study to Assess the Tolerance and Efficacy of DARATUMUMAB.
Brief Title: New Therapeutic Target for Toxic Epidermal Necrolysis (TEN) Using Anti-CD38+ Monoclonal Antibodies.
Acronym: NET-CD38
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); INSERM U1111 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL23_1000; 2024-512164-63-00 (EU CTIS Number); 2024-512164-63-00 (Other: UE Trial (CTIS) Number)
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Toxic Epidermal Necrolysis; Immunotherapy; Cutaneous Adverse Drug Reactions (CADR)
Keywords: Toxic Epidermal Necrolysis (TEN); Stevens-Johnson Syndrome (SJS); anti-CD38+; DARATUMUMAB; Simon design; Lyell syndrome
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, open-label phase I/II study using an optimal two-stage SIMON-type design for efficacy/tolerance evaluation (Simon, 1989), with an additional stage for tolerance evaluation alone... :
  1. After the first three inclusions, and two months of follow-up, a safety analysis with an opinion from the Independent Study Monitoring Board (DSMB) and an efficacy analysis (Simon's plan) will be carried out. If the rules allow (at least one patient with cessationof progression and a positive opinion from the DSMB concerning safety), 3 new patients will be included.
  2. After the first 6 inclusions and two months' follow-up, a safety analysis with a DSMB opinion will be carried out. If the DSMB opinion is favorable, 3 additional patients will be included.
  The 2-month follow-up period is sufficient for the collection of clinico-biological criteria of interest.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Single intravenous infusion of DARATUMUMAB 16 mg/kg body weight.
  Interventions: Drug: DARATUMUMAB (DARZALEX®)

INTERVENTIONS:
Drug: DARATUMUMAB (DARZALEX®) — A single injection of DARZALEX 16 mg/kg body weight administered by intravenous infusion (day 1) in addition to standard symptomatic treatment of NET until re-epidermalization.

SUMMARY:
Toxic Epidermal Necrolysis (TEN) are rare diseases that are dermatologic emergencies characterized by widespread epidermal necrosis and sloughing of skin. A hundred patients are affected each year in France. The main symptom is bullous and skin detachment > 10% which gradually progresses to extensive necrosis of the 100% BSA epidermis. The mortality rate is around 15-20% due to visceral inflammatory injuries and serious bacterial infections. The morbidity is also very important (92% at 1 year), especially ophthalmologic with high risk of blindness. There is currently no effective treatment.

Our team recently demonstrated that the severity of the disease correlates with the quantity and quality of CD8+ T lymphocytes which are activated in the active phase of disease. An activation marker has been identified, the CD38 receptor, which is very strongly expressed on the T clones responsible for the disease in the skin or blood of patients The CD38 receptor is the target of several commercial therapeutic antibodies, including DARATUMUMAB, which is currently used for the treatment of myeloma. DARATUMUMAB is a depleting antibody that eliminates cells strongly expressing this receptor.

The hypothesis is that a single intravenous infusion of DARATUMUMAB upon hospital admission of a patient with drug-induced NET would eliminate pathogenic T cells, thereby slowing disease progression, severity (% BSA with skin detachment, mortality rate) and sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Adult, over 18 years old, with drug-induced SJS/NET, proven or very strongly suspected (indirect argument of certainty) and confirmed by the evaluator.
* SJS or NET or overlap syndrome evolving for less than 7 days prior to inclusion and with a progression of the detachment or rash observed within 48 hours prior to DARATUMUMAB treatment.
* Negative hepatitis B screening (HBs, anti HBs and HBc).
* The patient (or a trusted support person, family member, or close relative in case of emergency) must be capable of understanding the objectives of the trial and must have given free, informed, and express consent.
* Patient affiliated to the Social Security system or benefiting from a similar system.
* Negative beta HCG pregnancy test for women of childbearing potential and agreement to use effective contraception during the study and up to 3 months after stopping DARATUMUMAB treatment.

Exclusion Criteria:

* Patient with Lyell syndrome induced by immunotherapy.
* Known hypersensitivity to the active substance (DARZALEX) or to one of the excipients (L-histidine, L-histidine hydrochloride monohydrate, L-methionine, Polysorbate 20 Sorbitol -E420).
* Patient with known hereditary fructose intolerance (HFI).
* Patient with known history of chronic obstructive pulmonary disease (COPD).
* Patient admitted with septic shock.
* PMNs < 1,500 /mm3 on CBC at inclusion visit.
* Pregnant or breast-feeding women.
* Patient under protective measures (safeguard, curatorship, guardianship) or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-10-29 (Estimated); Primary Completion 2028-10-29 (Estimated); Study Completion 2029-04-29 (Estimated)

PRIMARY OUTCOMES:
From baseline up to 24 hours after end of infusion: tolerance criteria defined as occurence of infusion related reactions, Cytokine release syndrome, main hemostasis parameters or variation in main biological parameters (blood ionogram). | At baseline and 24 hours after completion of the infusion of DARZALEX. If a clinical symptom or reaction is observed during infusion, an additional blood samples will be taken after a single intravenous infusion of DARZALEX 16 mg/kg body weight at day 1.
  Tolerance criteria according to NCI-CTCAE v5 criteria is defined as occurence of infusion related reactions; Cytokine release syndrome is characterized by increased levels of serum pro-inflammatory mediators; Main hemostasis parameters (prothrombin time (PT), activated partial thromboplastin time (APTT), fibrinogen (FBG), thromobin time (TT), and D-dimer (DD); Variation in main biological parameters (blood ionogram).
Efficacy defined as stop of disease progression at Day 6 | Day 6 after an intravenous injection of darzalex (16mg/kg)
  The cessation of disease progression at day 6 (D6) will be assessed by evaluating the change in the percentage of body surface area with skin detachment (detached and/or bullous surfaces, and/or associated with Nikolsky's sign) between the baseline (before daratumumab administration) and day 6 (D6), according to the following rules :
  * ≤ 2% for Stevens-Johnson Syndrome,
  * ≤ 5% for overlap syndrome
  * ≤ 10% for Lyell syndrome And without any new lesion with skin detachment. The percentage of body surface area with skin detachment will be evaluated based on the stable burn table using the E-Burn® application Day 6 after an intravenous injection of darzalex (16mg/kg) in addition to the reference symptomatic treatment (Day 1 = infusion of darzalex treatment)
The occurrence of grade 3 or higher cardiovascular, renal, thyroid, or intestinal adverse events within two months of injection (seven times the nine-day half-life of daratumumab) | Up to 2 months after the DARATUMUMAB infusion.
  Occurrence of grade >=3 cardiovascular, renal, thyroid or intestinal adverse events, according to NCI-CTCAE v5 criteria.

SECONDARY OUTCOMES:
Measure time between index date (onset of first symptom) and initiation of DARATUMUMAB treatment (Day 1) | From date of onset of first symptoms leading to the diagnosis of TEN (Toxic Epidermal Necrolysis) until the unique infusion of DARATUMUMAB treatment at (Day 1)]
  Total number of days between the unique intravenous infusion of DARATUMUMAB at day 1 and onset of first symptoms leading to the diagnosis of TEN (Toxic Epidermal Necrolysis)
Stop TEN progression delay: Time in days from start of DARATUMUMAB injection (Day 1) to cessation of progression | From the date of DARATUMUMAB infusion (Day 1) until the documented date of stopping progression of TEN, assessed up to 12 months or date of death from any cause
  Total number of days between intravenous infusion of DARATUMUMAB (day 1) and the documented stopping progression of TEN
Complete re-epidermalization delay: Time in days from start of DARATUMUMAB infusion (Day 1) to complete re-epidermalization | From the date of DARATUMUMAB infusion (day 1) until the documented date of complete re-epidermization, assessed up to 12 months or date of death from any cause.
  The complete re-epidermalization is defined as disappearance of skin erosions AND return to normal skin. The complete re-epidermalization is the total number of days between DARATUMUMAB injection (day 1) to complete re-epidermalization.
Hospital stay : measure the length of stay in one of the intensive care, burn, or internal medicine departments at Hôpital Édouard Herriot. | From admission to end of 12-month follow-up period
  Length of stay in E. Herriot hospital units care: Time between admission and discharge from E Herriot hospital
Co-morbidities associated with the NET: document ophthalmological, gynecological, pulmonary, digestive, psychiatric, urological, stomatological/ORL, dermatological, hepatic, nephrological sequelae at 2, 6 and 12 months after Day1 (injection of Darzalex). | At 2 months, 6 months and 12 months after Day 1 (injection of Daratumumab)
  Absence or presence of any co-morbitity: ophthalmological, gynecological, pulmonary, digestive, psychiatric, urological, stomatological/ORL, dermatological, hepatic and nephrological adverse event related to the disease and grade according to NCI-CTCAE v5 criteria.
Overall survival measure at Day 15 and 12 months after Darzalex infusion (D1) | At Day15 and 12 months after Darzalex infusion (Day 1).
  Overall survival rate defined as percentage of deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Reference Center for Toxic, Toxin and Toxidermal Bullous Dermatoses - E. Herriot Hospital, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided